CLINICAL TRIAL: NCT01917461
Title: Observational, Prospective Study to Evaluate Biomarkers as Indicators of Bacterial or Viral Infection During Acute Infectious Diseases
Brief Title: Observational, Prospective Clinical Study to Evaluate Biomarkers as Indicators of Acute Bacterial or Viral Infections
Acronym: CURIOSITY
Status: Completed | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MM-1001-BV
Record Dates: First submitted 2013-07-31; First posted 2013-08-06 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: LRTI; UTI; Gastroenteritis; Systemic Infections/Bacteremia/Meningitis; Fever Without Source
MeSH Terms: conditions — Gastroenteritis; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples Nasopharyngeal samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational prospective study of an in-vitro diagnostic (IVD) assay planned to enroll 632 subjects. The study will be conducted in two stages: Stage A is aimed at identifying individual biomarkers and constructing a multi-parametric diagnostic model, whereas Stage B is aimed at testing the multi-parametric diagnostic model using a fresh cohort of patients.

A collection of clinical, radiological and laboratory data will be gathered in order to establish a final diagnosis. Blood samples will be analyzed and the levels of approximately 700 and 250,000 biomarkers will be determined using immunoassays and molecular measurements respectively.

A final diagnosis will be determined based on a majority decision of a panel of three or more independent physicians. Based on the final diagnosis, the accuracy of individual biomarkers and combined sets of biomarkers for differentiating between distinct groups of patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients who are at least one month old and are willing (either the subject or his legal guardian) to sign an informed consent will be eligible for inclusion. For the infectious and non-infectious disease groups, additional inclusion criteria have to be met. These will include:

In the Infectious disease group:

* Peak fever >37.5°C (99.5°F)
* Clinical suspicion of an acute infectious disease
* Symptoms duration ≤ 12 days

In the Non-infectious disease control group:

- A non-infectious disease or healthy individuals

Exclusion Criteria:

Patients who will meet one or more of the following criteria will be excluded from the study:

* Evidence of another episode of acute infectious disease in the last two weeks
* Diagnosed congenital immune deficiency (CID)
* Current treatment with immunosuppressive therapy such as: Active chemotherapy,Post-transplant drugs,High dose steroids (>1 mg/kg/day prednisone or equivalent).
* Active radiotherapy
* Immune-modulating/suppressive drugs including monoclonal antibodies, intravenous immunoglobulin (IVIG), cyclosporine, and anti-TNF agents
* Current treatment with immune stimulants such as: Interleukin (IL)-2, Granulocyte-Monocytes/Granulocyte colony-stimulating factor (GM/G-CSF),Interferon.
* An active hematological malignancy
* A diagnosis of myelodysplastic syndrome or myeloproliferative disease
* A proven or suspected human immunodeficiency virus (HIV)-1, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects aged one month of age and older from both genders that attend the hospital or the emergency room (ER) due to a suspected acute infectious disease or due to a non-infectious disease (e.g. Trauma).
Sampling Method: Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of a multi-parametric diagnostic assay in differentiating between bacterial and viral etiology in patients with an acute infectious disease | 0-10 days after the initiation of symptoms
  We will evaluate the sensitivity and specificity of a multi-parametric diagnostic model, incorporating up to five different blood bio-markers in differentiating between bacterial and viral etiology in patients with an acute infectious disease.

SECONDARY OUTCOMES:
The sensitivity and specificity of individual biomarkers in differentiating between bacterial and viral etiology in patients with an acute infectious disease | 0-10 days after the initiation of symptoms
  We will evaluate the sensitivity and specificity of individual bio-markers in differentiating between bacterial and viral etiology in patients with an acute infectious disease.
The sensitivity and specificity of a multi-parametric assay in differentiating between mixed (bacterial and viral co-infection) and pure viral infections in patients with an acute infectious disease | 0-10 days after the initiation of symptoms
  We will evaluate the sensitivity and specificity of a multi-parametric diagnostic assay incorporating up to five different blood bio-markers, in differentiating between mixed infection(bacterial and viral co-infection) and pure viral infection in patients with an acute infectious disease.

CONTACTS AND LOCATIONS:
Overall Officials: Kfir Oved, Dr., Study Director — MeMed Diagnostics Ltd.
Locations (2):
- Israel (2):
  - Hillel Yaffe Hospital, Hadera, Israel
  - Bnei Zion Hospital, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No